CLINICAL TRIAL: NCT05873283
Title: Is Central Lymph Node Dissection Necessary in Suspected Papillary Thyroid Cancer and Papillary Thyroid Cancer?
Brief Title: Papillary Thyroid Cancer and Central Lymp Node Dissection
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20210310
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Papillary Thyroid Cancer
Keywords: papillary thyroid cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Papillary cancer is a disease that spreads through lymphatic ways and its treatment is surgery. We performed prophylactic central dissection in addition to bilateral total thyroidectomy in patients with bethesda 5 and bethesda 6 biopsy results. We evaluated the pathology results retrospectively.

ELIGIBILITY:
Inclusion Criteria:

- B5 and B6 biopsy results

Exclusion Criteria:

- lobectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with B5 and B6 biopsy results who underwent bilateral total thyroidectomy and central lymph node dissection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Reaching 100 patients was the first target | 18 months
  100 patients

CONTACTS AND LOCATIONS:
Locations (1):
- BasaksehirCamSakuraSehirH, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozel TM, Soytas Y, Akbulut S, Celik A, Yildiz G, Karatay H, Sari S. The necessity of prophylactic central lymph node dissection in clinically n0 papillary thyroid carcinoma: perspective from the endemic region. Langenbecks Arch Surg. 2025 Mar 28;410(1):109. doi: 10.1007/s00423-025-03667-y. PMID 40153045